CLINICAL TRIAL: NCT07272265
Title: The Effectiveness and Safety in High-risk Patients Receiving First-line Atezolizumab and Bevacizumab Combined With Hepatic Arterial Infusion Chemotherapy of FOLFOX for HCC: a Retrospective Study
Brief Title: The Effectiveness and Safety in High-risk Patients Receiving First-line Atezolizumab and Bevacizumab Combined With HAIC for HCC: a Retrospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAIC+TA Retrospective
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: FOLFOX-HAIC; Atezolizumab; Bevacizumab; high-risk HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOX+TA (Experimental): FOLOFOX-HAIC plus Atezolizumab and Bevacizumab
  Interventions: Drug: Atezolizumab & Bevacizumab; Procedure: FOLFOX-HAIC

INTERVENTIONS:
Drug: Atezolizumab & Bevacizumab — Atezolizumab 1200mg & Bevacizumab 15mg/kg Q3W
Procedure: FOLFOX-HAIC — hepatic artery infusion chemotherapy of oxaliplatin, leucovorin, and fluorouracil

SUMMARY:
This is a multicenter，retrospective study to explore the effectiveness and safety of Atezo/Bev plus hepatic artery infusion chemotherapy (HAIC) among adult patients with high-risk HCC in real-world clinical practice in China. Eligible patients diagnosed with high-risk HCC initiating the study treatment of interest between 28 October 2020 and 31 June 2025 will be included in this study. Secondary data from medical records of approximately 10 sites across China will be utilized.

ELIGIBILITY:
Inclusion criteria:

* Aged ≥ 18 years at the initiation of Atezo/Bev plus HAIC
* Initiating Atezo/Bev between 28 October 2020 and 31 June 2025
* Diagnosed with high-risk HCC as evidenced clinically or by radiology, histology or cytology before or at the initiation of Atezo/Bev plus HAIC. The evidence of being diagnosed as "high-risk" was based on the IMbrave 150, including any of the following:

  * tumor invasion of the main trunk or contralateral branch of the portal vein (Vp4)
  * bile duct invasion
  * tumor occupancy of 50% or more of the liver
* At least one visit record after the initiation of Atezo/Bev plus HAIC

Exclusion criteria:

* Diagnosed with concomitant cancer except for basal cell carcinoma before or at the initiation of Atezo/Bev plus HAIC
* Participating in interventional clinical studies before or at initiating Atezo/Bev plus HAIC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | 6 months
  defined as time from index date to death from any cause.

SECONDARY OUTCOMES:
Real-world progression-free survival (rwPFS) | 6 months
  defined as time from index date to the earlier of clinician-anchored progressive disease (may include but are not limited to local tumor progression, disease recurrence, new metastasis, or clinical progression anchored by clinicians) or death from any cause.
Time to discontinuation (TTD) | 6 months
  defined as time from the initiation to discontinuation of Atezo/Bev plus HAIC.
Time to next treatment (TTNT) | 6 months
  defined as time from the initiation of Atezo/Bev plus HAIC to the initiation of next systemic treatment.
Serum alpha-fetoprotein (AFP) reduction | 6 months
  defined as > 50% reduction in AFP level after 3 months (± 4 weeks) of the initiation of Atezo/Bev plus HAIC.
Prothrombin induced by the absence of vitamin K or antagonist- II (PIVKA-II) reduction | 6 months
  defined as > 50% reduction in PIVKA-II level after 3 months (± 4 weeks) of the initiation of Atezo/Bev plus HAIC.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 30 days
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China